CLINICAL TRIAL: NCT02414737
Title: Ovarian Stimulation Single Injection Elonva- The OSSIE Study
Brief Title: Ovarian Stimulation Single Injection Elonva
Acronym: OSSIE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Flinders Fertility (Industry)
Collaborators: Flinders University (Other)
Responsible Party: Principal Investigator, Professor Kelton Tremellen, Professor of Reproductive Medicine, Flinders Fertility
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AU/1/2 C8B110
Record Dates: First submitted 2015-04-08; First posted 2015-04-13 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- corifollitrophin alfa (Experimental): corifollitrophin alfa used as COH stimulant in IVF
  Interventions: Drug: corifollitrophin alfa

INTERVENTIONS:
Drug: corifollitrophin alfa — use of a single dose of corifollitrophin alfa to provide adequate controlled ovarian hyperstimulation during IVF treatment
  Other Names: Elonva

SUMMARY:
We would like to propose that it may be possible to use a solitary dose of Elonva (corifollitrophin alpha) as the sole gonadotrophin (FSH) stimulant for the vast majority of women undergoing IVF, assuming that it is possible that "coasting" (withholding short acting rFSH) from day 8 of the stimulation until trigger/ oocyte retrieval will still result in a significant number of mature oocytes being produced and an acceptable pregnancy rate.

DETAILED DESCRIPTION:
Elonva (corifollitrophin alfa) has been shown to be a very effective rFSH stimulant for Controlled Ovarian Hyperstimulation (COH) in the setting of IVF treatment. Its long duration of action (7 days) results in a significant reduction in the number of COH stimulation injections (average of 3 injections v 9 injections in the traditional "short acting" r FSH COH), with 30% of patients requiring only a single Elonva injection for their COH (Engage study, Devroey et al 2009). It is assumed that a reduction in the number of required COH injections will have the advantages of improved patient acceptability and better compliance due to a reduction in room for error. Despite these advantages the clinical uptake of Elonva has been slow due to 2 principal concerns among clinicians:

1. A tendency for Elonva COH to result in a higher ovarian response with increased risk of Ovarian Hyper-Stimulation Syndrome (OHSS). While this risk of OHSS was not statistically significant in the pivotal Engage study, there was still a numerically greater chance of OHSS and a greater chance of the IVF cycle being cancelled due to OHSS risk in the Elonva arm compared to the traditional Puregon arm. Since women at high risk of OHSS were excluded from the Engage study, clinicians perceive that the risk of OHSS is likely to be significantly greater in the more heterogeneous general clinical population. Whether this is a correct assumption is still up for debate, but it is a perceived issue with the existing Elonva protocol that must be addressed if Elonva is to become used widely as a COH stimulant.
2. According to the Engage and Ensure studies, the majority (70%) of women using Elonva require "top up"short acting Puregon rFSH, with an average of 2 doses being required before the patients reach the criteria for triggering and oocyte retrieval. As a result clinics are required to teach two different injection protocols, increasing the time required to educate the patient and possibly increasing the risk of confusion. The ability to deliver a solitary COH stimulant without the need for any "top up" Puregon would be a major advantage.

Rationale We would like to propose that it may be possible to use a solitary dose of Elonva as the sole COS rFSH stimulant for the vast majority of women undergoing IVF, assuming that it is possible that "coasting" (withholding short acting rFSH) from day 8 of the stimulation until trigger/ oocyte retrieval will still result in a significant number of mature oocytes being produced.

In the setting of OHSS it is common practice to withhold any further rFSH stimulant towards the end of the COS process. It is generally accepted that medium size follicles of 14 mm or greater will continue to develop to maturity in the absence of rFSH stimulation, while smaller follicles will regress. This has the therapeutic advantage of reducing estradiol levels and OHSS risk in women at high risk of OHSS. With this coasting physiology in mind, we propose that provided a single injection of Elonva can result in a significant number of follicles being 14 mm or greater by day 8 of stimulation, further rFSH will not be required. Results from the Engage study (Doody et al 2011) reveal that by day 8 of stimulation on average there were 5.1 follicles of 15 mm or greater. Therefore even if no further "top up" rFSH was given from day 8, one could expect to get at least 5 mature oocytes from an oocyte retrieval triggered by hCG in the next 2 days. While 5 mature oocytes is significantly less than what was produced by the traditional Elonva protocol using additional rFSH (average 10.8 in the Engage study, 10.7 in the Ensure study), this could be perceived as a significant advantage since it will likely result in a significant reduction in OHSS risk, a perceived problem with the traditional Elonva protocol. If we assume a 70% fertilization rate and that approximately half of all embryos are of good quality by day 4/5 of culture, the production of > 3 mature oocytes should ensure the generation of at least one good quality embryo for transfer with a good chance of pregnancy. This type of low impact stimulation is likely to be very popular in Europe and Australia where clinicians already accept the benefits of mild COS.

In summary, if we are able to provide evidence in this pilot study that a single injection of Elonva can result in the majority of women reaching oocyte retrieval with the production of at least 3 mature oocytes, while giving good fresh embryo transfer pregnancy rates and no OHSS, the coasting Elonva protocol may become a significant clinical protocol for low impact COS in the future.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing a GnRH antagonist cycle of IVF as part of their personal fertility treatment
* Eligible for the use of the 150 mcg dose of Elonva according to Australian PBS requirements (weight > 60 kg, antral follicle count < 20)
* Intention of undergoing a fresh embryo transfer.
* No major sperm quality issues (ejaculate sperm concentration > 5 million/ ml, motility > 25% neat sample). ICSI for the indication of poor morphology would be acceptable for trial enrollment.
* Maternal age 18-37 years inclusive.

Exclusion Criteria:

* Low ovarian reserve (antral follicle count 2-10 mm < 7, early follicular phase FSH > 10 IU/L, < 4 oocytes prior IVF cycle on a dose of rFSH > 150 IU).
* Ovarian pathology (PCOS, ovarian cyst, endometrioma, poor trans-vaginal ultrasound ovary access).
* 2 or more previous cycles of IVF (stimulated cycles) in which a live birth pregnancy did not result, or one prior stimulated cycle of IVF and 2 or more frozen embryo transfer cycles without a live birth outcome (possible implantation failure).
* Significant pelvic pathology likely to impair embryo implantation (fibroids, polyps, uterine septum, hydrosalpinx).
* Intention to freeze all embryos with nil fresh transfer (pre-implantation genetic screening, oncology fertility preservation).
* Known renal impairment
* Use of a long down regulation or "flare" IVF protocol.

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-02; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Oocyte maturity - number of mature oocytes (metaphase II oocytes) retrieved in IVF cycle | IVF cycle (2 weeks approximately)
  number of mature oocytes (metaphase II oocytes) retrieved in IVF cycle

OTHER OUTCOMES:
cryopreservation of embryos - number of good quality embryos available for cryopreservation | IVF cycle
  number of good quality embryos available for cryopreservation

CONTACTS AND LOCATIONS:
Overall Officials: Kelton Tremellen, MD PhD, Principal Investigator — Flinders University
Locations (1):
- Flinders Fertility, Bedford Park, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No